CLINICAL TRIAL: NCT05644028
Title: A Pilot Study of a Blended Intervention Targeting Emotion Dysregulation in Adults with ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 494659
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Emotion regulation Intervention (Experimental): An 8-week blended intervention targeting emotion dysregulation in ADHD
  Interventions: Behavioral: Emotion Regulation Intervention for ADHD

INTERVENTIONS:
Behavioral: Emotion Regulation Intervention for ADHD — The intervention will be based on principles from dialectic behavioral therapy. The overall aim of the intervention is to improve emotion regulation skills. The intervention will consist of eight face-to-face group sessions and a digital companion app that the participants can use to practice skills between the sessions. The groups will include mindfulness-based exercises, homework review, introduction to new skills, and peer discussions.

SUMMARY:
The current study aims to investigate the feasibility and preliminary clinical effects of a blended psychological intervention targeting emotion dysregulation in adults with ADHD.

DETAILED DESCRIPTION:
Adults with ADHD with co-occurring deficits in emotion regulation are expected to have more severe impairment than those without such deficits in several life domains. Both pharmacological and psychological treatment interventions for adults with ADHD tend to target core symptoms of inattention and hyperactivity, and there are few available interventions targeting emotional symptoms. The current study aims to investigate the feasibility and preliminary clinical effects of a blended psychological intervention targeting emotion dysregulation in ADHD. The intervention consists of eight face-to-face group sessions and a companion app to be used by the participants between the sessions for skills training. The investigators seek to recruit between 15 to 20 adults with ADHD to participate in the pilot study. Feasibility outcomes include adherence, treatment satisfaction and treatment credibility. Self-report questionnaires assessing emotion dysregulation, ADHD symptoms, quality of life, anxiety and depression will be used to examine preliminary clinical effects. There will also be conducted qualitative process interviews to examine the participants expectations and experiences with the program. The investigators expect the intervention to be feasible and to find positive preliminary effects. The findings from the study will be of importance for to further improve the intervention for for a future randomized-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. A diagnosis of ADHD
3. Current problems with emotion regulation as indicated with a score above 80 on the Difficulties in Emotion Regulation Scale (DERS)
4. Access to a smartphone

Exclusion Criteria:

1. Current self-reported diagnosis of severe psychiatric illness such as ongoing substance abuse or psychosis.
2. High risk of suicidality, as indicated by a) has attempted suicide within the last year, b) has previously attempted suicide and reports suicidal ideation, or c) reports current ideations and has a plan or preferred method.
3. Other ongoing psychological treatment for ADHD or other psychiatric illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
The Credibility and Expectancy Questionnaire (CEQ) | Up to 12 weeks
  The third item from the The Credibility and Expectancy Questionnaire (CEQ) will be used to assess treatment credibility. The third item states "How confident would you be in recommending this treatment to a friend with similar challenges? The item is rated on a scale from 1 (none at all confident) to 9 (very confident)
Open questions on treatment satisfaction | Up to 12 weeks
  At the post-intervention assessment, the participants will be asked whether they are likely to continue using the exercises from the intervention in the future and whether they have experienced any adverse events, where the participants will have the option to elaborate in an open text-field. There will also be conducted qualitative interviews with the participants to examine their experiences (positive and negative) with the program.
Treatment adherence | Up to 12 weeks
  Number of attended group sessions and number of completed homework assignments

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | Up to 12 weeks
  The measure is a self-report questionnaire that is commonly used to assess emotion dysregulation in clinical populations. The scale includes 36 items rated on a 5-point scale ranging from "Never" (1) to "Almost always" (5), yielding a total score of between 36 - 180, where a higher score indicate a higher degree of emotion dysregulation.
The Adult ADHD Self-Rating Scale (ASRS) | Up to 12 weeks
  The scale assesses symptoms of inattention (nine items), and symptoms of hyperactivity-impulsivity (nine items) and includes a total of 18 items. The response type consists of a 5-point scale with options "Never" (0), "Rarely" (1), "Sometimes" (2), "Often" (3) or "Very Often" (4) giving the scale a maximum score of 72 for full-scale ASRS and 36 on each of the two subscales of inattention and hyperactivity-impulsivity. A higher score indicate a higher severity in symptoms.
The Adult ADHD Quality of Life Measure (AAQoL) | Up to 12 weeks
  The measure assesses quality of life during the past two weeks and is specifically developed for adults with ADHD. The scale comprises 29 items rated on a scale from "Not at all/Never" (1) to "Extremely/Very Often" (5), yielding a total score between 0 - 100 points. The scale also included four subscales: life productivity, psychological health, life outlook, and relationships, all yielding a score between 0 - 100 points. A higher score indicates better quality of life.
Hospital Anxiety and Depression Scale (HADS) | Up to 12 weeks
  The scale examine symptoms of depression and anxiety. The scale consists of 14 items with response options ranging from 0-3, with 3 being the most severe level of symptoms. The scale yields one total score, ranging from 0-42, and one subscale score from depression, and one subscale for anxiety, ranging from 0-21.
The Behavior Rating Inventory of Executive Functioning Adult version (BRIEF-A) | Up to 12 weeks
  The Behavior Rating Inventory of Executive Functioning Adult version (BRIEF-A) is a self-report questionnaire assessing executive functioning in everyday life. The scale consists of 75 items and are rates on a 3-point scale from "Never" (1) to "Often" (3).

CONTACTS AND LOCATIONS:
Overall Officials: Astri Lundervold, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nordby ES, Guribye F, Schonning V, Andersen SL, Kuntsi J, Lundervold AJ. A Blended Intervention Targeting Emotion Dysregulation in Adults With Attention-Deficit/Hyperactivity Disorder: Development and Feasibility Study. JMIR Form Res. 2024 Jan 17;8:e53931. doi: 10.2196/53931. PMID 38231536
- [Background] Nordby ES, Schonning V, Barnes A, Denyer H, Kuntsi J, Lundervold AJ, Guribye F. Experiences of change following a blended intervention for adults with ADHD and emotion dysregulation: a qualitative interview study. BMC Psychiatry. 2025 Jan 20;25(1):56. doi: 10.1186/s12888-025-06476-1. PMID 39833731